CLINICAL TRIAL: NCT06981403
Title: The Effect of the Virtual Escape Room Method on Pediatric Drug Administration in Nursing Students:
Brief Title: The Effect of the Virtual Escape Room Method on Pediatric Drug Administration Knowledge, Self-Efficacy, Clinical Comfort, and Anxiety in Nursing Students: A Randomized Controlled Study
Acronym: Pediatric Drug
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SU
Record Dates: First submitted 2025-04-21; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Medication
Keywords: Virtual escape room, nursing, paediatric drug administration, self-efficacy, anxiety, clinical comfort
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Intervention: virtual escape room game education and control: standard education
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): virtual escape room game-based pediatric medication management education
  Interventions: Behavioral: virtual escape room game-based pediatric medication management education
- control group (No Intervention): standard education

INTERVENTIONS:
Behavioral: virtual escape room game-based pediatric medication management education — 3 period aplied virtual escape room game-based pediatric medication management education
  Arms: intervention group

SUMMARY:
Children are particularly vulnerable to injuries resulting from medication errors due to the severity of the illness, the need for high-risk drugs with a narrow therapeutic range, and the frequent use of intravenous infusions. Despite recent advances in pharmacological research in the pediatric population, the issue of availability of medications suitable for children has not yet been resolved. Therefore, in the pediatric group, it is necessary to calculate the correct dosage of medications, prepare them with appropriate methods, and dilute them with suitable diluents. The literature indicates that dosage calculation errors are the most common medication errors in neonatal and pediatric patients. It is unclear whether nursing students are adequately prepared to provide pharmaceutical care in practice. Nursing students and new nursing graduates often lack the competence to administer medications safely. Therefore, training should be planned to enhance students' competencies and knowledge levels. The inclusion of newer methods in educational techniques has become essential as technology and social media increasingly engage nursing students. Today's nursing students need alternative, innovative ways to be involved in the learning process. Among these methods, gaming is used in nursing education to support the development of critical thinking and practical skills in students. Game-based learning has the potential to engage students and enhance learning, offering numerous advantages alongside innovation and excitement. In light of these advantages, the aim of this study is to evaluate the effects of a virtual escape room application on nursing students' knowledge level, self-efficacy, clinical comfort, and anxiety in pediatric medication management.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd year nursing student,
* Having a computer or smart phone,
* Volunteering to participate in the study

Exclusion Criteria:

* Students who repeated a grade,
* Students who suspended their nursing education,
* Students who cancelled their registration

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Pediatric Medication Management Knowledge Level Form | pre-test (before the game education initiative), post-test (after the game education initiative) and follow-up (after 6 months)
  It is a form consisting of 31 questions to measure the knowledge level of students about pediatric drug administration. Students will be asked to mark the true or false option in this form. Opinions of expert academicians and nurses in the field were taken for the prepared information questions.
Pediatric Nursing Student Clinical Comfort and Worry Assessment Tool | pre-test (before the game education initiative), post-test (after the game education initiative) and follow-up (after 6 months)
  pediatricNursing Student Clinical Comfort and Worry Assessment Tool was developed by Al-Qaaydeh and Lassche Macintosh in 2012 to determine the areas of concern and comfort of nursing students who were first in the pediatric clinic in the clinical environment (Al-Qaaydeh et al, 2012). The Turkish validity and reliability study of the scale was conducted by Arslan et al in 2018. The scale consists of a total of 11 questions, 6 of which are used to determine the comfort level of students during the pediatric clinic and 5 of which are used to determine the anxiety level. This measurement tool is a 4-point Likert-type scale. The scale options include "1-Strongly agree", "2- Agree", "3- Disagree" and "4-Strongly disagree". The scale has reverse coded questions. The 3rd and 5th items of the comfort sub-dimension of the scale are reverse items, therefore the items were scored in reverse. Cronbach alpha reliability value was found to be 0.68 for the Comfort Level and 0.89 for the Anxiety sub-d
Self-Efficacy Scale for Medication Administration in Children for Nursing Students | pre-test (before the game education initiative), post-test (after the game education initiative) and follow-up (after 6 months)
  The Self-Efficacy Scale for Medication Administration in Children for Nursing Students was developed by Bektaş et al in 2021. The scale consists of 16 items and two sub-dimensions. It is a 5-point Likert type and is 1=Absolutely inadequate, 2=Somewhat adequate, 3=Partially adequate, 4=Adequate, 5=Absolutely adequate. The lowest score obtained from the scale is 16 and the highest score is 80. The scale has no cut-off point, as the score increases, the students' self-efficacy regarding pediatric medication administration increases. The scale does not have a reverse-scored item. The Cronbach's alpha coefficient for the entire scale was .94, .91 for the first medication preparation sub-dimension, and .87 for the second medication administration sub-dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No